CLINICAL TRIAL: NCT05311163
Title: MITRA-EF: A Multi-Center Registry Evaluating Left Ventricular Function in Patients Undergoing Transcatheter Mitral Edge-To-Edge Repair
Brief Title: Change in LVEF Following Transcatheter Mitral Edge-To-Edge Repair
Acronym: MITRA-EF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RMC-18-0352
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: MitraClip — Transcatheter Mitral Edge-To-Edge Repair

SUMMARY:
Little is known regarding the impact of transcatheter mitral valve edge-to-edge repair (TEER) on the acute changes in left ventricular ejection fraction (LVEF) and the effect of an acute reduction in LVEF, the so-called "afterload mismatch" (AM), on prognosis.

We thereby aim to assess changes in LVEF after TEER, identify rate and predictors AM, and estimate its impact on prognosis.

DETAILED DESCRIPTION:
Following surgical mitral valve repair for primary mitral regurgitation (MR), improved left ventricular (LV) and left atrial remodeling was demonstrated. However, little is known regarding the impact of percutaneous mitral edge-to-edge repair in patients with secondary MR or those with primary MR who are not candidates for surgery. Studies in these populations are limited, vary in the inclusion criteria and the etiology of mitral regurgitation. Some show no improvement in LV ejection function (LVEF) following percutaneous repair despite reduced LV end-diastolic diameter (LVEDD) and LV end-systolic diameter (LVESD), whereas in others an improvement in LVEF was shown. One study suggests reverse remodeling only in patients with lower values of logistic EuroSCORE and STS scores, LV end-diastolic volume index (LVEDVi), right ventricular end systolic area, and pulmonary artery systolic pressure (PAPs) at baseline evaluation and in multivariate analysis, only PAPs remained an independent predictor of improvement. Another study utilizing cardiovascular magnetic resonance to assess extent and predictors of reverse remodeling (defined by reduction of LVEDVi>15% compared to baseline) demonstrated improvement in only 34% of the patients, predicted by improvement in MR volume and MR fraction. In the landmark Cardiovascular Outcomes Assessment of the MitraClip Percutaneous Therapy for Heart Failure Patients With Functional Mitral Regurgitation (The COAPT Trial), LVEF had deteriorated following both repair and the control arm of medical therapy alone, albeit at a lower rate in patients treated with the MitraClip device (reduction of 5.6±1.2% versus 8.8±1.1%, p=0.048).

It was shown, in a few preliminary trials, that a significant number of patients undergoing transcatheter mitral edge-to-edge repair suffer from an acute reduction in left ventricular function. This so called "afterload mismatch" resulted in worsened prognosis in this patient population, as compared with controls.

Nevertheless, the information available in the current literature is limited and based on relatively smaller studies. We therefore wish to learn more about patients undergoing transcatheter mitral edge-to-edge repair, encompassing both primary and secondary mitral regurgitation, assess dynamics in left ventricular function during and after the admission, identify predictors of an acute reduction in left ventricular function and understand its impact on prognosis.

In this international, multicenter registry, consecutive patients undergoing TEER are included. We aim to assess changes in LVEF and LV end-diastolic volume (LVEDV) immediately after the procedure. We will then assess rates of AM, defined as a reduction of >15% in LVEF or an increase of >15% in LVEDV, its impact on all-cause mortality, MACE (composite end point of all-cause death, surgery and grade 3+ or 4+ mitral regurgitation) and LVEF at 12 months, as well as predictors for AM.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* patients who are taken immediately to surgery following the procedure
* those who did not have echocardiographic information in the first 30 days post TEER
* patients who have undergone combined mitral and tricuspid repair
* severe non-cardiovascular diseases such as systemic infection or malignancy
* cardiogenic shock presenting at baseline

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing TEER using the MitraClip percutaneous mitral valve repair (Abbott Vascular, Inc., Santa Clara, California) are included.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 12 months
  Rates of all cause death
MACE | 12 months
  Rates of major adverse cardiac events (MACE= a composite of death, need for mitral surgery or percutaneous repair and rates of grade 3+ or 4+ mitral regurgitation)

SECONDARY OUTCOMES:
LV Function and size | 12 months
  12-month LVEF and LVEDV
NYHA | 12 months
  New York Heart Association (NYHA) classification
Heart failure admissions | 12 months
  Number of heart failure admissions
Need for mitral surgery or percutaneous repair | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Central District, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perl L, Kheifets M, Guido A, Agricola E, Denti P, Wild MG, Praz F, Rubbio AP, Bedogni F, De Marco F, Beeri R, Shuvy M, Melillo F, Montorfano M, Freixa X, de la Fuente Mancera JC, Giordano A, Finizio F, Van Mieghem NM, Ooms JFW, Fam N, O'Connor C, Toggweiler S, Levi A, Shapira Y, Schwartzenberg S, Pidello S, D'Ascenzo F, Angelini F, Haberman D, Crimi G, Porto I, Cozzi O, Giannini F, Tarantini G, Maisano F, Kornowski R; MITRA-EF study *. Acute Reduction in Left Ventricular Function Following Transcatheter Mitral Edge-to-Edge Repair. J Am Heart Assoc. 2023 Jul 4;12(13):e029735. doi: 10.1161/JAHA.123.029735. Epub 2023 Jun 22. PMID 37345813